CLINICAL TRIAL: NCT07288814
Title: A Single-Arm, Open-Label Ib/II Study of Mitoxantrone Hydrochloride Liposome and Enlonstobart Combination Treatment in Patients With Relapsed or Refractory Peripheral T Cell Lymphoma（PTCL）
Brief Title: Mitoxantrone Hydrochloride Liposome and Enlonstobart Combination Treatment in Patients With Relapsed or Refractory Peripheral T Cell Lymphoma (PTCL)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yet-Sen University Cancer Center (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Huiqiang Huang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Sun Yet-Sen University Cancer Center
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-PTCL-K08
Record Dates: First submitted 2025-11-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Peripheral T Cell Lymphoma
Keywords: Mitoxantrone Hydrochloride Liposome; Enlonstobart
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone hydrochloride liposome combined with enlonstobart (Experimental)
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome & Enlonstobart

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome & Enlonstobart — Mitoxantrone hydrochloride liposome: ①Phase Ib：16 mg/m2、20 mg/m2 ，D1，q4w; ②Phase II：RP2D, D1，q4w, Up to 6 cycles
  Enlonstobart: 360mg，D1，q4w (The maintenance treatment phase is q3w), Up to 1 year

SUMMARY:
To evaluate the safety of mitoxantrone hydrochloride liposome combined with enlonstobart in the treatment of relapsed or refractory peripheral T-cell lymphoma, to determine the optimal dosage of mitoxantrone hydrochloride liposome within the combination regimen, and to assess the efficacy of the combined therapy.

DETAILED DESCRIPTION:
This is a single-arm, phase Ib/II study to investigate the safety and efficacy of mitoxantrone hydrochloride liposome combined with enlonstobart in the treatment of relapsed and refractory peripheral T-cell lymphoma, and the optimal dose of mitoxantrone hydrochloride liposome. In the dose-escalation phase, the initial dose of mitoxantrone hydrochloride liposome injection was 16mg/m2, and two dose groups of 16mg/m2, 20 mg/m2, D1, q4w were designed. Enlonstobart was administered at a fixed dose of 360mg, D1, q4w. Dose-limiting toxicity (DLT) was assessed after cycle 1. Six cycles of induction therapy were planned. After induction therapy, if the response evaluation was CR/PR, maintenance treatment with enlonstobart (360mg, D1, q3w) could be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Centrally confirmed histopathological/cytologic diagnosis of PTCL with the following subtypes:

   1. Peripheral T-cell lymphoma, not otherwise specified (PTCL, NOS);
   2. Systemic anaplastic large cell lymphoma (ALK+ and ALK-);
   3. Follicular helper T (TFH) cell lymphoma of lymph nodes, including angioimmunoblastic, follicular, NOS;
   4. and any other PTCL subtypes deemed by the investigator to be eligible for inclusion.
2. Voluntary participation in clinical study; Fully understand and informed the study and sign the written informed consent;
3. Age ≥18 years old, and ≤ 75 years old, regardless of gender;
4. Met the criteria of relapsed/refractory lymphoma: Relapsed lymphoma was defined as relapsed lymphoma more than 6 months after achieving complete remission (CR) after initial chemotherapy. Refractory lymphoma was defined as any of the following criteria: 1) tumor shrinkage < 50% or disease progression after at least 4 courses of standard chemotherapy; 2) achieved CR with standard chemotherapy, but relapsed within half a year;
5. ECOG performance status score: 0-2;
6. Expected survival time ≥3 months;
7. There must be at least one measurable or evaluable lesion that meets the Lugano 2014 criteria for lymphoma:

1)Measurable lesion: Nodal lesions with major diameter greater than 1.5cm and minor diameter greater than 1.0cm as assessed by PET/CT or Computed Tomography (CT) and/or Magnetic Resonance Imaging (MRI); Or the length of extranodal lesions >1.0cm; 2)Evaluable lesions: PET-CT showed increased uptake in lymph nodes or extranodal regions (higher than liver) and imaging features consistent with lymphoma; 8.Have adequate organ and bone marrow function, defined as follows:

1. Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L(≥1.0×109/L in patients with bone marrow involvement); platelet count (PLT) ≥ 75×109/L(≥50×109/L in patients with bone marrow involvement), hemoglobin (HGB) ≥ 8.0 g/dL; The patients had not received granulocyte growth factor, platelet transfusion, or red blood cell transfusion within 14 days before the examination;
2. Liver function: serum total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN, liver invasion ≤3.0×ULN); alanine aminotransferase (ALT) and aspartate transferase (AST) ≤2.5×ULN (liver invasion ≤5.0×ULN);
3. Renal function: serum creatinine (Cr) ≤1.5×ULN.
4. Coagulation function: International Normalized Ratio (INR) ≤1.5 × ULN; Prothrombin Time (PT), Activated PartialThromboplastin Time (APTT) ≤1.5×ULN (unless the subject is receiving anticoagulant therapy, And PT and APTT at screening were within the expected range for anticoagulant therapy).
5. Thyroid stimulating hormone (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) within the normal range ±10% (Note: non-autoimmune causes of abnormal TSH, FT3 and FT4 can be maintained in the normal range after replacement treatment of hypothyroidism can be enrolled).

   9.Patients who had received previous antineoplastic therapy could not be enrolled until the toxicity of previous treatment returned to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade score ≤1 or the baseline level; 10.Women of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose of medication; Effective contraception should be used from the time of informed consent until 6 months after the last dose of study drug.

Exclusion Criteria:

1. Patients with hemophagocytic lymphohistiocytosis;
2. Patients with active infection or with obvious B symptoms and high fever should be excluded according to the comprehensive judgment of the investigators;
3. The subject's previous history of antineoplastic therapy meets one of the following conditions:

   1. Failure to achieve CR or PR after previous treatment with mitoxantrone or mitoxantrone liposome, or relapse within 6 months after treatment;
   2. Prior treatment with anthracyclines or anthraquinones and cumulative dose of doxorubicin > 550 mg/m2 (liposomal doxorubicin > 2000 mg/m2, epirubicin > 1000 mg/m2, pirarubicin > 1000 mg/m2, mitoxantrone > 160 mg/m2);
   3. Received anti-tumor treatment (including chemotherapy, targeted therapy, traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received clinical trial drugs within 4 weeks or 5 half-lives (whichever came first) before the first use of the study drug;
   4. patients who received autologous hematopoietic stem-cell transplantation or allogeneic hematopoietic stem-cell transplantation within 100 days of the first dose of treatment;
4. Hypersensitivity reaction to any study drug or its components;
5. Patients with known allergy to any component of the monoclonal antibody;
6. Patients with a known history of Human Immunodeficiency Virus (HIV) infection and/or acquired immunodeficiency syndrome;
7. Patients with active chronic hepatitis B or active hepatitis C. Hepatitis B SurfaceAntigen (HBsAg) or hepatitis B core Antibody (HBcAb) or Hepatitis C Virus (HCV) during the screening period HCV) antibody positive patients must be further tested for Hepatitis B Virus (HBV) DNA (no more than 1000 copies /mL or 500 IU/mL) and HCV RNA (no more than the lower limit of detection of the assay), Enrollment in the trial occurred after the exclusion of patients with active hepatitis B or hepatitis C infection requiring treatment. Hepatitis B virus (HBV) carriers, medically stable hepatitis B (DNA > 1000 copies /mL or 500IU/mL) and cured hepatitis C patients are eligible for enrollment.
8. Cardiac function and disease is one of the following:

   1. long QTc syndrome or QTc interval >480 ms;
   2. complete left bundle branch block, degree II or III atrioventricular block;
   3. severe, uncontrolled arrhythmia requiring medical treatment;
   4. New York College of Cardiology grade ≥ III;
   5. cardiac ejection fraction (LVEF) less than 50%;
   6. a history of myocardial infarction, unstable angina, major unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities within 6 months before recruitment;
9. Receive live attenuated vaccine (except influenza vaccine) within 4 weeks before enrollment or during the study period;
10. Previous or current concurrent cancer (except for effectively controlled non-melanoma basal cell carcinoma of the skin, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the previous five years);
11. Those with central nervous system involvement;
12. Lactating women;
13. Subjects receiving systemic glucocorticoid therapy or other immunosuppressive therapy for a condition within 14 days before starting study treatment (topical, ocular, intra-articular, nasal, and inhaled glucocorticoids were allowed (minimal systemic absorption); Short-term (≤ 7 days) use of glucocorticoids was permitted for preventive treatment (e.g., contrast allergy) or for the treatment of nonautoimmune conditions (e.g., delayed hypersensitivity from contact allergens).
14. Had undergone major surgery within 28 days before starting study treatment, or had undergone radiation therapy within the previous 90 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose limited toxicities (DLTs) | Cycle 1 (28 days)
  Adverse events (AE) defined as DLT events per protocol
Phase Ib: Recommended Phase II Dose (RP2D) | through Phase Ib study completion, an average of 3 months
  RP2D based on Phase Ib results
Phase II: Objective response rate (ORR) | Up to 1 years
  Response is assessed according to the 2014 lugano criteria

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 1 years
  Response is assessed according to the 2014 lugano criteria
Disease control rate (DCR) | Up to 1 years
  Response is assessed according to the 2014 lugano criteria
Progression-free survival（PFS） | Up to 2 years
  From the time subjects were enrolled to the time of disease progression (in any way) or death from any cause.
Overall survival (OS) | Up to 2 years
  From the date of inclusion to date of death, irrespective of cause.
Adverse events(AE) | From the first day of medication to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard. Hematologic and non-hematologic toxicity.

IPD SHARING:
Plan to Share IPD: No